CLINICAL TRIAL: NCT06979999
Title: The Effects of Positive End-Expiratory Pressure (PEEP) on Optic Nerve Sheath Diameter (ONSD) in Patients Undergoing Laparoscopic Cholecystectomy Under General Anesthesia: A Prospective Interventional Study
Brief Title: The Effects of Positive End-expiratory Pressure (PEEP) on Optic Nerve Sheath Diameter in Laparoscopic Cholecystectomy
Acronym: PEEPON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Seval KILBASANLI, Asst. Prof., Nigde Omer Halisdemir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/54; 2024/54 (Other: Niğde Ömer Halisdemir University Faculty of Medicine)
Record Dates: First submitted 2025-04-29; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Positive End-expiratory Pressure (PEEP); Intracranial Pressure; Optic Nerve Sheath Diameter; Mechanical Ventilation
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP Group (Experimental): This arm includes patients undergoing laparoscopic cholecystectomy under general anesthesia. All participants receive 10 cmH₂O PEEP after pneumoperitoneum creation, and optic nerve sheath diameter (ONSD) is measured intraoperatively at predefined time points.
  Interventions: Procedure: Positive End-Expiratory Pressure (PEEP)

INTERVENTIONS:
Procedure: Positive End-Expiratory Pressure (PEEP) — Application of 10 cmH₂O PEEP during mechanical ventilation after pneumoperitoneum creation in patients undergoing laparoscopic cholecystectomy.

SUMMARY:
This prospective interventional study will evaluate the effects of applying positive end-expiratory pressure (PEEP) at 10 cmH₂O on optic nerve sheath diameter (ONSD) in patients undergoing elective laparoscopic cholecystectomy under general anesthesia. A total of approximately 80 adult patients (ASA physical status I-III) will be included following informed consent.

ONSD will be measured using a high-frequency linear ultrasound probe at three predefined intraoperative time points: (T0) 10 minutes after initiation of mechanical ventilation, (T1) 10 minutes after pneumoperitoneum creation, and (T2) 30 minutes after pneumoperitoneum creation. Dynamic lung compliance, peak airway pressure (Ppeak), end-tidal CO₂ (EtCO₂), heart rate, mean arterial pressure, and SpO₂ will also be recorded.

The aim is to assess whether the application of PEEP influences intracranial pressure indicators, particularly ONSD, during laparoscopic procedures. The study may provide valuable insights into the neurophysiological effects of intra-abdominal pressure and mechanical ventilation strategies in surgical patients.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (age ≥ 18 years)

American Society of Anesthesiologists (ASA) physical status I-III

Scheduled for elective laparoscopic cholecystectomy under general anesthesia

Signed informed consent

Exclusion Criteria:

* resence of acute or chronic eye disease

Uncontrolled hypertension

Asthma or known chronic pulmonary disease

Any neurological disorders

Body mass index (BMI) > 35 kg/m²

Use of medications known to affect intracranial pressure

Refusal to participate after signing informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-05-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Change in Optic Nerve Sheath Diameter (ONSD) | Intraoperative; T0, T1, T2
  ONSD will be measured via ultrasound at 3 time points during surgery.

SECONDARY OUTCOMES:
Change in Peak Airway Pressure (Ppeak) | Intraoperative measurement at T0, T1, and T2
  Peak airway pressure will be measured using the ventilator settings at three predefined intraoperative time points to evaluate respiratory mechanics during PEEP application.
Change in Dynamic Lung Compliance | Intraoperative measurement at T0, T1, and T2
  Dynamic lung compliance will be calculated using the formula: Tidal Volume / (Ppeak - PEEP) and measured at three intraoperative time points.
Change in End-Tidal Carbon Dioxide (EtCO₂) | Intraoperative measurement at T0, T1, and T2
  End-tidal CO₂ levels will be recorded intraoperatively to monitor changes in ventilation efficiency during surgery.
Changes in Heart Rate (HR) and Mean Arterial Pressure (MAP) Time Frame | Intraoperative measurement at T0, T1, and T2
  Heart rate and mean arterial pressure will be recorded at predefined time points to assess hemodynamic stability during surgery.
Peripheral Oxygen Saturation (SpO₂) | Intraoperative continuous monitoring and recorded at T0, T1, and T2
  Peripheral oxygen saturation will be monitored continuously and recorded at specified intraoperative time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Training and Research Hospital, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No